CLINICAL TRIAL: NCT03301363
Title: Simultaneous Or Sequential multiPoint Pacing in Cardiac Resynchronization Therapy
Brief Title: Simultaneous or Sequential Multipoint Pacing
Acronym: SCOPE-CRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, Chief of Arrhythmology Department IRCCS SAn Donato Policlinico, University of Milan, Italy, IRCCS Policlinico S. Donato
Other Study IDs: SCOPE-CRT IRCCSDonato
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CRT — Subjects scheduled to be implanted for CRT by a Quadripolar Pacing System

SUMMARY:
The purpose of this study is to compare electrical acute changes between simultaneous and sequential LV pacing and to assess the paced QRSd over a range of inter- and intra-ventricular programmable delays setting during MPP pacing.

DETAILED DESCRIPTION:
The study will be a prospective, single-arm, non-randomized, non-blinded, acute study conducted at CRT device implant and prior to subject discharge. Subjects scheduled to be implanted with a Quadripolar Pacing System who provide informed consent will undergo "Enrollment" and participate in "SCOPE-CRT" study. Enrollment and device implant can occur in the same day. Including Enrollment, each subject's participation is expected to be 1-2 days. The total duration of the study is expected to be 12 months, including Enrollment. Enrollment will include the Informed Consent process, physical examination, and collection of demographics, cardiovascular history, medical history, and medications.

During CRT implant, surface ECG and PV loop recordings will be taken over the different programmable MPP settings. Following data collection, CRT device programming will be left to the discretion of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with approved indication for CRT by European Society of Cardiology/European Heart Rhythm Association guidelines (ESC/EHRA)
* QRS duration > 130 ms
* Ability to provide informed consent for study participation
* At least 18 years of age

Exclusion Criteria:

* Myocardial infarction within 40 days before enrolment

  * NYHA Class IV
  * Tachyarrhythmia caused by temporary or reversible irritation, e.g. poisoning, electrolyte imbalance, hypoxia, sepsis or acute myocardial infarction
  * Such frequent VT or VF that the therapies would cause an unacceptably rapid depletion of the device batteries
  * VT with few or without clinically relevant symptoms
  * VT or VF treatable by surgery
  * Concomitant diseases that would substantially limit a positive prognosis
  * Accelerated intrinsic rhythm
  * Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 selected heart failure patients with approved indication for CRT by European Society of Cardiology/European Heart Rhythm Association guidelines (ESC/EHRA) will be enrolled for this prospective study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute QRS duration changes during multipoint CRT | 1 day during CRT
  Quantify acute changes in surface ECG QRS duration between simultaneous and sequential LV pacing during MPP pacing.

SECONDARY OUTCOMES:
Acute ECG QRS duration changes during multipoint CRT | 1 day during CRT
  Quantify acute changes in surface ECG QRSd over a range of inter- and intra-ventricular programmable delays setting during multipoint CRT pacing.
  •
Acute changes in hemodynamics between simultaneous and sequential LV pacing during multipoint CRT | 1 day during CRT
  Quantify acute changes in hemodynamics between simultaneous and sequential LV pacing during multipoint CRT pacing over a range of inter- and intra-ventricular programmable delays settings.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — IRCCS San Donato University Hospital Policlinico San Donato, Milan, Italy
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No